CLINICAL TRIAL: NCT02034565
Title: Study of Bioavailability of Apixaban Solution Formulation Relative to Apixaban Tablets in Healthy Subjects
Brief Title: Phase 1 Bioavailability Study of Apixaban Solution Formulation Relative to Apixaban Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-029
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: Apixaban tablet (Experimental): Apixaban Film coated Tablet Single dose 10 mg orally
  Interventions: Drug: Apixaban
- Treatment B: Apixaban oral solution (Experimental): Apixaban Solution Single dose 10 mg orally
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: BMS - 562247

SUMMARY:
The purpose of this study is to assess the oral bioavailability of Apixaban solution formulation (Treatment B, 10 mg as 25 mL x 0.4 mg/mL) relative to Apixaban tablets (Treatment A, 10 mg as 2 x 5 mg tablets) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Any significant acute or chronic medical illness or relevant trauma (e.g., history of chronic hypertension, bacterial endocarditis, hemorrhagic stroke, motor vehicle accident resulting in significant head trauma or internal injuries)
* History or evidence of abnormal bleeding or coagulation disorder (e.g., easy bruising or gingival bleeding, prolonged bleeding after dental extraction, postpartum, or after trauma, wounds or surgery)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services, Neptune City, New Jersey, United States

REFERENCES:
- [Result] Song Y, Wang X, Perlstein I, Wang J, Badawy S, Frost C, LaCreta F. Relative Bioavailability of Apixaban Solution or Crushed Tablet Formulations Administered by Mouth or Nasogastric Tube in Healthy Subjects. Clin Ther. 2015 Aug;37(8):1703-12. doi: 10.1016/j.clinthera.2015.05.497. Epub 2015 Jul 15. PMID 26188837
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 participants were enrolled; 14 were randomized and treated. Reasons for non-randomization include 23 no longer met study criteria, 4 withdrew consent, 6 due to study being full, and 1 completed an alternate treatment. 13 participants completed the study.
Groups:
- Treatment A, Then Treatment B; Treatment B, Then Treatment A: Each participant was given two interventions, one per period, with a 4 day washout in between periods.
  Treatment A: Single dose apixaban film-coated tablet, 10 milligrams (mg) via 2 x 5 mg tablets, administered orally
  Treatment B: Single dose apixaban solution, 10 milligrams (mg) via 25 milliliters (mL) x 0.4 mg/mL, administered orally
Period: Overall Study
Arm/Group | Treatment A, Then Treatment B | Treatment B, Then Treatment A
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- All Treatment Groups: All Randomized Participants
Arm/Group | All Treatment Groups
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 36 [28 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean of the Maximum Observed Plasma Concentration (Cmax) of Apixaban
Description: Serial blood samples for pharmacokinetic analysis were collected at selected times up to 72 hours after each dose. Maximum observed plasma concentration (Cmax) is measured in nanograms per milliliter (ng/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose per intervention
Population: All treated participants with available pharmacokinetic (pk) data
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Treatment A: Apixaban Tablet: Single dose apixaban 10 mg (film-coated tablet) administered orally
- Treatment B: Apixaban Oral Solution: Single dose apixaban 10 mg (solution) administered orally
Arm/Group | Treatment A: Apixaban Tablet | Treatment B: Apixaban Oral Solution
Number analyzed (Participants) | 14 | 13
ng/mL | 293.994 [245.998 to 351.354] | 287.164 [242.331 to 340.291]
Statistical Analysis 1: Comparison: Treatment A: Apixaban Tablet vs Treatment B: Apixaban Oral Solution; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.977, 90% CI 2-sided [0.756 to 1.261]

2. Primary Outcome: Adjusted Geometric Mean of the Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero Extrapolated to Infinite Time AUC(INF) of Apixaban
Description: Serial blood samples for pharmacokinetic analysis were collected at selected times up to 72 hours after each dose. AUC(INF) is measured in nanogram hours per milliliter (ng*h/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose per intervention
Population: All treated participants with available pk data
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A: Apixaban Tablet | Treatment B: Apixaban Oral Solution
Number analyzed (Participants) | 13 | 13
ng*h/mL | 2712.477 [2414.339 to 3047.432] | 2848.968 [2557.946 to 3173.101]
Statistical Analysis 1: Comparison: Treatment A: Apixaban Tablet vs Treatment B: Apixaban Oral Solution; Test type: Superiority or Other; Ratio of adjusted geometric means = 1.050, 90% CI 2-sided [0.938 to 1.176]

3. Primary Outcome: Adjusted Geometric Mean of the Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] of Apixaban
Description: Serial blood samples for pharmacokinetic analysis were collected at selected times up to 72 hours after each dose. AUC(0-T) is measured in nanogram hours per milliliter (ng*h/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose per intervention
Population: All treated participants with available pk data
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A: Apixaban Tablet | Treatment B: Apixaban Oral Solution
Number analyzed (Participants) | 13 | 13
ng*h/mL | 2668.310 [2372.198 to 3001.385] | 2784.366 [2497.506 to 3104.175]
Statistical Analysis 1: Comparison: Treatment A: Apixaban Tablet vs Treatment B: Apixaban Oral Solution; Test type: Superiority or Other; Ratio of adjusted geometric means = 1.043, 90% CI 2-sided [0.933 to 1.167]

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment-Related Adverse Events (AEs), Deaths or Discontinuation of Study Drug Due to AEs
Description: AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during the study and up to 28 days past study discontinuation. The select AEs were determined using the Medical Dictionary for Regulatory Activities (MedDRA, v13).
Time Frame: Day 1 to 30 days after last dose of study drug
Population: All treated participants
Measure: Number; unit: participants
Groups:
- Arm A: Apixaban Tablet: Single dose apixaban 10 mg (film-coated tablet) administered orally
- Arm B: Apixaban Oral Solution: Single dose apixaban 10 mg (solution) administered orally
Arm/Group | Arm A: Apixaban Tablet | Arm B: Apixaban Oral Solution
Number analyzed (Participants) | 14 | 13
participants
  SAE | 0 | 0
  Treatment-Related AE | 0 | 1
  Deaths | 0 | 0
  Treatment-Related Deaths | 0 | 0
  Discontinuation of Study Drug Due to AEs | 1 | 0

5. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Clinical laboratory tests were performed pre-study and at selected times throughout the study. Marked laboratory abnormalities were defined as laboratory assessments meeting the following investigator-specified criteria: Leukocytes < 0.9* lower limits of normal (LLN), absolute neutrophils + bands <= 1.500 10*3 cells/microliter, white blood cells (WBC) urine value >= 2+. These laboratory abnormalities were not considered clinically significant and therefore not adverse events.
Time Frame: Pre-study screen (Day -1) to Day 8 or day of study discharge
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Arm A: Apixaban Tablet | Arm B: Apixaban Oral Solution
Number analyzed (Participants) | 14 | 13
participants
  Leukocytes, Low | 1 | 1
  Absolute Neutrophils + Bands, Low | 1 | 1
  WBC, Urine, High | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 30 days
Arm/Group | Arm A: Apixaban Tablet | Arm B: Apixaban Oral Solution
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 4/14 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Apixaban Tablet (N=14) | Arm B: Apixaban Oral Solution (N=13)
Constipation (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less